CLINICAL TRIAL: NCT05663359
Title: Randomized Comparative Study With Two Wavelengths 1470 nm and 1940 nm for the Treatment of Varicose Veins of the Lower Limbs by Endovenous Laser.
Brief Title: Study on Treatment of Varicose Veins by Endovenous Laser (1940 nm vs 1470 nm)
Acronym: NEWWAVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Pasteur (Other)
Responsible Party: Principal Investigator, Nicolas NEAUME, Principal Investigator, MD, Clinique Pasteur
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A01722-41
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Varicose Veins
Keywords: Endovenous laser ablation (EVLA)
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1940 nm (Active Comparator): Endovenous laser at 1940 nm
  Interventions: Procedure: EVLA 1940 nm
- 1470 nm (Active Comparator): Endovenous laser at 1470 nm
  Interventions: Procedure: EVLA 1470 nm

INTERVENTIONS:
Procedure: EVLA 1940 nm — Treatment of varicose veins by endothermic ablation with an endovenous laser at 1940 nm
  Arms: 1940 nm
Procedure: EVLA 1470 nm — Treatment of varicose veins by endothermic ablation with an endovenous laser at 1470 nm
  Arms: 1470 nm

SUMMARY:
The goal of this clinical trial is to compare efficacy of two wavelength for EndoVenous Laser Ablation (EVLA) in treatment of varicose veins of the lower limbs.

The main questions it aims to answers are :

1. Is the increase of wavelength form 1470 nm to 1940 nm affect the efficacy of varicose veins treatment ?
2. Is the increase of wavelength reduce complication or pain ? Participants are patients with varicose veins of lower limbs and candidate for endovenous laser ablation.

After laser ablation patients will be followed during 5 years for clinical evaluation, recording potential treatment complications and quality of life evaluation.

Researchers will compare strategy 1(EVLA with an endovenous laser at 1940 nm) vs strategy 2 (EVLA with an endovenous laser at 1470 nm) in varicose veins treatment to see if efficacy of treatment is not reduce, and to see if complications of EVLA treatment can be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Primary insufficiency of the great saphenous vein (GSV) and/or small saphenous vein (SSV)
* Patient candidate for endothermic treatment of the lower limbs
* CEAP: C2 - C6
* Patient with a target vein diameter (GSV and/or SSV) >= 3 mm throughout the target vein segment
* Patient affiliated or beneficiary of a social security scheme
* Patient having signed the informed consent

Exclusion Criteria:

* Patient with a current serious pathology and/or a life expectancy of less than 5 years
* Patient who has had a deep or superficial vein thrombosis in the previous 6 months
* Obliterating arteriopathy of the lower limb concerned, with an IPS < 0.8 or > 1.3
* Patient with post-thrombotic obstructive syndrome at the popliteal and/or femoral and/or iliac stage on the ipsilateral lower limb
* Patient with primary or post-thrombotic axial deep venous reflux on the ipsilateral lower limb
* Suspicion of non-post-thrombotic iliac compression on echo-doppler
* Contraindication to the planned treatment technique
* Patient whose geographical distance is not compatible with the follow-up of the study
* Pregnant or breastfeeding women
* Patient linguistically or psychologically unable to understand the information given, to give informed consent or to answer the study questionnaires.
* Protected patients: Adults under guardianship, or other legal protection; Hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2031-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Anatomical success | At 5 years
  Closure of the target vein

SECONDARY OUTCOMES:
VAS Pain | Day 0, Day 8, Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  Visual Analogue Scale (0-100 mm); higher is worse
Adverse Events | Day 0, Day 8, Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  Adverse events related to endovenous treatment
Venous Clinical Severity | Day 0, Day 8, Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  Venous Clinical Severity Score (VCSS) ; score between 0 to 30; higher is worse
Symptoms | Day 0, Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  VEINES Sym (VEnous INsufficiency Epidemiologic and Economic Study - Symptoms) questionnaire
Patient quality of life (1) | Day 0, Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  VEINES Sym (VEnous INsufficiency Epidemiologic and Economic Study - quality of life ) questionnaire
Patient quality of life (2) | Day 0, Month 6, Year 1, Year 2, Year 3, Year 4, Year 5
  EuroQol-5 Dimension (EQ5D) Quality of life survey

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas NEAUME, MD, Principal Investigator — Clinique Pasteur
Locations (1):
- Clinique Pasteur, Toulouse, France